CLINICAL TRIAL: NCT03988829
Title: Strategic Training to Optimize Neurocognitive Functions in Older Adults
Acronym: ViCTOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas at Dallas (Other)
Collaborators: University of Texas Southwestern Medical Center (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IRB 20-06; 1R56AG060052-01 (NIH)
Record Dates: First submitted 2019-05-10; First posted 2019-06-18 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2020-11

CONDITIONS: Cognitive Aging; Functional Magnetic Resonance Imaging
Keywords: randomized control trial; cognitive training; simulation games; improving brain function; improving cognition; functional magnetic resonance imaging

STUDY DESIGN:
Intervention Model Description: We will conduct a randomized control trial on healthy older adults, where attentional control demands in cognitive training will be systematically increased using engaging game-based simulations. There are three parallel arms: predictable low attentional control (Arm 1: Low-C), unpredictable high attentional control (Arm 2: High-C), and a commercially-available strategy video game (Arm 3: High-C+). In all three training arms, neural and cognitive changes in both near and far tasks will be examined immediately after the 8-week long intervention. Long-term cognitive changes will also be assessed at 6 months after completion of training. The far and near cognitive outcomes that will be examined are episodic memory (the primary cognitive outcome) and executive control (the secondary cognitive outcome).
  Additionally, a single-session functional neuroimaging dataset will be collected in a functional control group of younger adults; they will not undergo any intervention.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: If a volunteer meets the inclusion and exclusion criteria, he or she will be randomized into one of the three training arms. This assignment will be based on a random computerized allocation plan, where the average cognitive frailty, age, education and gender distribution will be maintained to be equivalent across the three arms. To maintain the balance between the arms, we will randomize between blocks of 15 participants. By randomly assigning participants in the training arms and by assessing outcomes by blinded experimenters, we will avoid selection bias and outcome assessment bias.
  No masking is required for the younger adults, as they will not be undergoing any training.
  The PI will be blinded to training assignment of any subject, and will only analyze de-identified data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low-C (Active Comparator): In an experimenter-designed simulation game, participants will be trained on predictable low attentional control shifts during working memory.
  Interventions: Behavioral: Low-C
- High-C (Experimental): In an experimenter-designed simulation game, participants will be trained on unpredictable high attentional control shifts during working memory.
  Interventions: Behavioral: High-C
- High-C+ (Experimental): In this commercially-available video game, in addition to unpredictable shifts of attentional control in working memory, task switching and resource planning will be trained.
  Interventions: Behavioral: High-C+

INTERVENTIONS:
Behavioral: Low-C — This is the active control group, where participants will be trained to play an experimenter developed game that requires least attentional control among all arms.
  Other Names: Predictable Bird Watch
  Arms: Low-C
Behavioral: High-C — In this intervention, participants will be trained on this experimenter developed game which requires a lot of attentional control.
  Other Names: Unpredictable Bird Watch
  Arms: High-C
Behavioral: High-C+ — A commercial video game will be used that requires a lot of demand on attentional control.
  Other Names: Video Game
  Arms: High-C+

SUMMARY:
The goal of the present randomized control trial is to evaluate the efficacy of a novel cognitive training approach using simulated games, where older adults will learn to flexibly deploy attentional control during working memory, for prevention of Alzheimer's Disease (AD). Based on our extensive pilot work, we expect training-related enhancements in both neural and cognitive functions on a broad range of cognitive abilities due to the importance of attentional control and working memory in many types of cognition. These outcomes are widely applicable to the cognitive health and the quality of life of elderly Americans, and have further potential to offset degenerative processes common to normal aging.

DETAILED DESCRIPTION:
Almost all older adults experience cognitive frailty with age, with around one-third of adults aged 85 or older suffering from Alzheimer's disease (AD). Cognitive frailty, particularly AD, threatens to overwhelm medical resources in the United States and much of the developed world. Therefore, it is important that we learn how to optimize and maintain cognitive performance in cognitively-frail older adults, particularly those who are at high risk of suffering from AD, such as adults over 70 years of age where more than half express AD pathology. The present multi-arm randomized control trial takes a novel theory-driven approach to enhancing cognition in older adults by training them to flexibly deploy attentional focus in working memory. Flexibility in allocating and switching attentional resources will be trained by having participants respond to unpredictable cues in working memory. The ability to flexibly and efficiently allocate attentional control underlies successful performance on a broad array of cognitive tasks. Hence, training in this area may enhance performance not only on related tasks (near transfer) but also on tasks that are perceptibly not related to the training task (far transfer).

The current proposal has three training arms and utilizes game-based simulations in all arms in healthy older adults. The first two arms use experimenter-designed simulation games, where participants will be trained on either predictable low attentional control (Arm 1) or unpredictable high attentional control (Arm 2) working memory games. The third arm uses a commercially available strategy game requiring the highest level of attentional control, by adding multi-tasking to the unpredictable attentional shifts in working memory. In all three training arms, neural and cognitive changes in near (secondary outcome) and far (primary outcome) transfer tasks will be examined immediately after the intervention; cognitive changes will also be assessed at 6-month post-training duration. Additionally, a single-session, baseline neuroimaging data (no training) will be collected in a functional control group of younger adults. We expect that the high attentional control training arms will greatly improve both near and far cognition in older adults, with cognitive frailty interacting with the extent to which attentional control is trained. High attentional control training arms are also expected to heighten compensatory brain activation after the intervention, for both near and far in-scanner transfer tasks, mimicking the baseline activity of younger brains. These training arms are also expected to positively impact brain structures that progressively decline with aging. This clinical trial will result in the development of behavioral intervention tools, which will have the potential to delay the onset of memory-related disorders, such as AD, by instantiating durable improvements in cognitive functions in older adults. Such interventions can not only improve an individual's quality of life but also decrease the financial burden of a rapidly aging society.

ELIGIBILITY:
Inclusion Criteria:

* At least a 10th grade education
* Learned English before age 5
* If female, not pregnant or likely to be pregnant
* Right-handed
* Mini Mental State (MMSE) score of 26 or greater (for older adults only), Montreal Cognitive Assessment (MoCA) score of 24 or more (for older adults only)
* The physical and sensory capacity sufficient to undertake a functional magnetic resonance imaging study

Exclusion Criteria:

* Color blindness assessed by the Ishihara Test for Color Deficiency
* Visual acuity of less than 20/30 on the Snellen eye chart after correction
* Diagnosis of any major psychiatric or neurologic disorders
* History of cardiovascular disease other than treated hypertension
* Illness or trauma affecting the central nervous system
* Substance/alcohol abuse, and medication with anti-depressants, anti-psychotics, or hypnotics other than occasionally at bedtime
* Structural magnetic resonance imaging reveal evidence of pathology (e.g. infarction)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2018-09-30 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Immediate Change in the Composite Score of Episodic Memory | 9-10 weeks (includes baseline assessment, training, and post-training assessment)
  Change in composite score of episodic memory from baseline to post-training (i.e., after 8 weeks of training). The composite score of episodic memory will include correct responses from 3 episodic memory tasks:
  1. Picture Sequence Memory
  2. Rey Auditory Verbal Learning Test (RAVLT)
  3. Story Recall (MMSE)
  For all tasks, alternative forms will be used for baseline testing and for post-training. Details of the tasks are listed below:
  1. Participants are asked to reproduce a sequence of pictures that is shown on the screen.
  2. Fifteen words are read to participants. Immediately after, the participant is asked to recall the entire list. This is repeated a few times.
  3. A short story is read to participant. Immediately after, the participant is asked to repeat the story.
6-month Change in the Composite Score of Episodic Memory | 8 months (=6 mo of retention + 9-10 weeks)
  Change in composite score of episodic memory from baseline to 6-months after completion of training (i.e., after 8 weeks of training). The composite score of episodic memory will include correct responses from 3 episodic memory tasks:
  1. Picture Sequence Memory
  2. RAVLT
  3. Story Recall (MMSE)

SECONDARY OUTCOMES:
Immediate Change in the Composite Score of Executive Control | 9-10 weeks (includes baseline assessment, training, and post-training assessment)
  Change in composite score of episodic memory from baseline to post-training (i.e., after 8 weeks of training). The composite score of executive control will include correct responses from 6 tasks:
  1. Task Switching Response Time (RT)
  2. Dimensional Change Accuracy
  3. Flanker RT
  4. Stroop RT
  5. Visual N-back RT
  6. Verbal Memory Updating Accuracy
  For all tasks, alternative forms will be used for baseline testing and for post-training.
6-month Change in the Composite Score of Executive Control | 8 months (=6 mo of retention + 9-10 weeks)
  Change in composite score of executive control from baseline to 6-months after completion of training (i.e., after 8 weeks of training). The composite score of executive control will include correct responses from 6 tasks:
  1. Task Switching RT
  2. Dimensional Change Accuracy
  3. Flanker RT
  4. Stroop RT
  5. Visual N-back RT
  6. Verbal Memory Updating Accuracy
  Alternate forms will be used at baseline and at 6-months after completion of training.

OTHER OUTCOMES:
Immediate Change in the Composite Score of Reasoning | 9-10 weeks (includes baseline assessment, training, and post-training assessment)
  Change in composite score of Reasoning from baseline to post-training (i.e., after 8 weeks of training). The composite score of reasoning will include correct responses from 2 tasks:
  1. Matrix Reasoning
  2. Visual Puzzle
  For all tasks, alternative forms will be used for baseline testing and for post-training.
Immediate Change in the Composite Score of Working Memory Capacity | 9-10 weeks (includes baseline assessment, training, and post-training assessment)
  Change in composite score of Working Memory Capacity from baseline to post-training (i.e., after 8 weeks of training). The composite score of working memory capacity will include correct responses from 2 tasks:
  1. List Sorting Working Memory
  2. Complex Span
  For all tasks, alternative forms will be used for baseline testing and for post-training.
6-month Change in the Composite Score of Reasoning | 8 months (=6 mo of retention + 9-10 weeks)
  Change in composite score of Reasoning from baseline to 6-months after completion of training (i.e., after 8 weeks of training). The composite score of reasoning will include correct responses from 2 tasks:
  1. Matrix Reasoning
  2. Visual Puzzle
  For all tasks, alternative forms will be used for baseline testing and at 6-months after completion of training.
6-month Change in the Composite Score of Working Memory Capacity | 8 months (=6 mo of retention + 9-10 weeks)
  Change in composite score of Working Memory Capacity from baseline to 6-months after completion of training (i.e., after 8 weeks of training). The composite score of working memory capacity will include correct responses from 2 tasks:
  1. List Sorting Working Memory
  2. Complex Span
  For all tasks, alternative forms will be used for baseline testing and at 6-months after completion of training.
Immediate Change in the Composite Score of Psychosocial Functioning - MIDUS-II | 9-10 weeks (includes baseline assessment, training, and post-training assessment)
  Change in composite score of Psychosocial Functioning from baseline to post-training (i.e., after 8 weeks of training). The composite score of psychosocial functioning will include correct responses from 4 tasks:
  1. MIDUS-II
  2. Cognitive Reserve Index
  3. Rivermead Behavioral Memory Test - III
  4. New general Self-efficacy Scale
  For all tasks, alternative forms will be used for baseline testing and for post-training.
6-month Change in the Composite Score of Psychosocial Functioning - MIDUS-II | 8 months (=6 mo of retention + 9-10 weeks)
  Change in composite score of Psychosocial Functioning from baseline to 6-months after completion of training (i.e., after 8 weeks of training). The composite score of psychosocial functioning will include correct responses from 4 tasks:
  1. MIDUS-II
  2. Cognitive Reserve Index
  3. Rivermead Behavioral Memory Test - III
  4. New general Self-efficacy Scale
  For all tasks, alternative forms will be used for baseline testing and at 6-months after completion of training.
Immediate Change in Processing Speed | 9-10 weeks (includes baseline assessment, training, and post-training assessment)
  Change in numbers of items correctly coded within 2 minutes on the Digit Symbol Substitution task from baseline to post-training (i.e., after 8 weeks of training).
  Alternative forms will be used for baseline testing and for post-training.
6-month Change in Processing Speed | 8 months (=6 mo of retention + 9-10 weeks)
  Change in numbers of items correctly coded within 2 minutes on the Digit Symbol Substitution task from baseline to post-training (i.e., after 8 weeks of training).
  Alternative forms will be used for baseline testing and at 6-months after completion of training.

CONTACTS AND LOCATIONS:
Overall Officials: Chandramallika Basak, PhD, Principal Investigator — The University of Texas at Dallas
Locations (1):
- The Center for Vital Longevity (UT Dallas), Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2019-02-20): https://cdn.clinicaltrials.gov/large-docs/29/NCT03988829/Prot_SAP_000.pdf
  • Informed Consent Form: Older adults (2019-01-25): https://cdn.clinicaltrials.gov/large-docs/29/NCT03988829/ICF_001.pdf
  • Informed Consent Form: Younger adults (2019-01-25): https://cdn.clinicaltrials.gov/large-docs/29/NCT03988829/ICF_002.pdf